CLINICAL TRIAL: NCT04419935
Title: Prognostic Impact of the Kind of Lymphadenectomy and Lymph Node Characteristics on Node-positive Patients Underwent Anatomical Lung Resection With or Without Adjuvant Therapy for Non-Small Cell Lung Cancer
Brief Title: Lymphadenectomy in NSCLC With and Without Adjuvant Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Chiappetta marco, Medical Doctor - Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3100
Record Dates: First submitted 2020-05-15; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: NSCLC; Lymph Node Metastases
Keywords: Thoracic Surgery; Adjuvant therapy
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Lymph Node Excision; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lymphadenectomy — Lymphadenctomy according with ESTS guidelines
  Other Names: adjuvant therapy

SUMMARY:
Adjuvant therapy in patients affected by NSCLC is indicated in surgically treated cases of N2 disease, while the actual guidelines reported the possibility of a case-by-case decision in case of N1 involvement.

On the other hand, the actual categorization of patients based on the hilar or mediastinal involvement (N1 or N2) risks to be too ineffective and straightforward for prognosis prediction and an indication of adjuvant treatments. This issue was underlined in the 8th TNM proposal for the N sub-classification, with a final proposal of different subgroups based on the number of involved stations. However, the IASLC committee noted that this proposal presented some limits due overlapping or not statistical significance among some survival curves, so the proposal was not adopted in the staging system. Moreover, the committee stated that the lack of information regarding some data such as the number of the resected or the metastatic nodes might affect the results and limited other proposals.

The objectives of this study are:

* To evaluate the prognostic role of the kind of lymphadenectomy, the number of the resected and/or metastatic lymph nodes in surgically treated N positive patients in terms of survival.
* To evaluate the indication and the role of adjuvant treatments in these patients.
* To identify patients with increased risk of early recurrence or poor survival based on the lymph node involvement characteristics In particular, data will be collect in a prospective database including clinical and pathological data, kind of lymphadenectomy, number of resected nodes, number of metastatic nodes, kind and schedule of adjuvant therapy and follow-up status

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age >18 years
* Non-Small Cell Lung Cancer Histology
* Anatomical lung resection (segmentectomy, lobectomy or bilobectomy, pneumonectomy)
* Pre-operative CT and PET evaluation
* Preoperative and postoperative tumour board discussion
* Intraoperative lymph node assessment (minimum 3 mediastinal stations harvested)
* Lymph node metastases

Exclusion Criteria:

* AGE < 18 years
* Pregnancy
* Psychiatric disease
* Wedge resection
* Distant metastases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients affected by Non-Small Cell Lung Cancer underwent surgical treatment with anatomical resection + lymphadenectomy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the prognostic role of the number of resected and metastatic lymph nodes in pathologically node-positive NSCLC patients underwent surgical resection | 5 years
  overall survival will be used to assess the prognostic role of number of resected and metastatic nodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Chiappetta, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided